CLINICAL TRIAL: NCT02314520
Title: Complications Associated With Central Venous Access in the NSICU: PICC vs CVC
Acronym: NSPVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Chris Zacko, Assistant Professor of Neurosurgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000582
Record Dates: First submitted 2014-11-26; First posted 2014-12-11 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: PICC; Central Venous Catheter; Central Line; Neuro ICU; Neuroscience ICU; CVC
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PICC (Active Comparator): Patients randomly assigned to receive a peripherally inserted central catheter and they will be monitored for either having a complication or no complication.
  Interventions: Device: peripherally inserted central catheter
- CVC (Active Comparator): Patients randomly assigned to receive a centrally inserted central catheter and they will be monitored for either having a complication or no complication.
  Interventions: Device: centrally inserted central catheter

INTERVENTIONS:
Device: peripherally inserted central catheter — Any complication associated with central access
  Arms: PICC
Device: centrally inserted central catheter — Central access not associated with any complication
  Arms: CVC

SUMMARY:
The goal of this study is to determine whether Peripherally Inserted Central Catheter or Centrally Inserted Venous Catheters have lower complication rates in the Neuroscience Intensive Care Unit. After admission to the Neuroscience ICU and if they require central access, patients will be randomized to receive a PICC or CVC and complications (such as pneumothorax, deep venous thrombosis, infection, etc.) will be tracked and compared between the two interventions.

ELIGIBILITY:
Inclusion Criteria:

Adult patients admitted to the NSICU, who require central access for the treatment of their illness.

Exclusion Criteria:

1. Current or recent (within 1 month) diagnosis of bacteremia
2. Current or recent (within 1 year with confirmed resolution by imaging) deep venous thrombosis
3. Existing central access
4. Non-English speaking
5. Requirement for emergent central access and unable to obtain consent in an emergency setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Central Line: Patients randomly assigned to receive a centrally inserted central catheter and they will be monitored for either having a complication or no complication.
  centrally inserted central catheter: Central access not associated with any complication
Period: Overall Study
Arm/Group | PICC | Central Line
Started | 72 | 80
Completed | 72 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PICC | Central Line | Total
Number analyzed (Participants) | 72 | 80 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (18) | 63.3 (13.6) | 61.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 35 | 45 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 80 | 152
Glasgow Coma Scale (Total) [Median (Standard Deviation); unit: points] — The Glasgow Goma Scale (GCS) gives a description of level of consciousness. Patients are assigned a minimum of 1 and maximum of 6 units on a scale for motor skills, a minimum of 1 and maximum of 5 units on a scale for verbal skills, a minimum of 1 and maximum of 4 units on a scale for eye opening function. The total GCS is a simple sum of all of the units on a scale with a minimum of 3 and maximum of 15. Higher values indicate higher neurologic function.
  points | 9.5 (4.0) | 10 (3.6) | 10 (3.8)
Hemiparesis [Count of Participants; unit: Participants] | 38 | 38 | 76
Diagnosis [Count of Participants; unit: Participants]
  stroke | 28 | 29 | 57
  subarachnoid hemorrhage | 14 | 18 | 32
  traumatic brain injury | 11 | 8 | 19
  intraparenchymal hematoma | 10 | 12 | 22
  myasthenia gravis | 0 | 1 | 1
  intraventricular hemorrhage | 0 | 1 | 1
  other | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Participants With Complications With Central Access Including Insertion
Description: Aggregation of all complications associated with central access including insertion
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PICC | Central Line
Number analyzed (Participants) | 72 | 80
Participants | 14 | 10
Statistical Analysis 1: Comparison: PICC vs Central Line; Test type: Superiority; p = 0.271, Fisher Exact — 0.05 is the threshold for significance for this primary outcome

2. Secondary Outcome: Number of Participants With Deep Venous Thrombosis
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PICC | Central Line
Number analyzed (Participants) | 72 | 80
Participants | 4 | 0

3. Secondary Outcome: Number of Patients With Complications Related to Insertion
Description: Any complication of insertion including technical failure
Time Frame: From the time of insertion until first confirmatory chest X-ray
Measure: Count of Participants; unit: Participants
Arm/Group | PICC | Central Line
Number analyzed (Participants) | 72 | 80
Participants | 8 | 6

4. Secondary Outcome: Number of Participants With a Central Line Associated Blood Stream Infection
Description: A Central access associated infection (CLABSI)
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PICC | Central Line
Number analyzed (Participants) | 72 | 80
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 Months
Description: Definitions do not differ.
Arm/Group | PICC | Central Line
All-Cause Mortality (participants affected / at risk) | 13/72 | 9/80
Serious Adverse Events (participants affected / at risk) | 4/72 | 1/80
Other Adverse Events (participants affected / at risk) | 0/72 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICC (N=72) | Central Line (N=80)
Deep venous thrombosis (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No